CLINICAL TRIAL: NCT03094676
Title: Effects of Massage as a Recuperative Technique in Different Moments of Application on Autonomic Cardiac Modulation and Cardiorespiratory Parameters
Brief Title: Effects of Massage in Different Moments of Application on Autonomic Cardiac Modulation and Cardiorespiratory Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Nilton Mantovani Junior, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 57584116.6.0000.5402
Record Dates: First submitted 2017-02-21; First posted 2017-03-29 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
Keywords: Massage; Autonomic nervous system; Recovery of Physiological Function; Heart Rate
MeSH Terms: interventions — Massage; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and the assessor will not receive information about the participant, not knowing, from which group the participant has just arrived for intervention in the investigator's case and the assessor will not receive group information in the HRV data packet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): Only the HRV will be followed for two hours without intervention.
- Only Massage (Experimental): Only the massage, and will have the monitoring of the HRV on the techniques and accompanied for two hours.
  Interventions: Other: Massage
- Only Exercise (Experimental): Only the exercise, and will have the monitoring of the HRV on the techniques and accompanied for two hours.
  Interventions: Other: Exercise
- Exercise and Massage immediately (Experimental): Performing the exercise and massage immediately after, will be accompanied by the HRV during the techniques and two hours after.
  Interventions: Other: Massage; Other: Exercise
- Exercise and Massage after recovery (Experimental): Performing the exercise and massage will be applicated after recovery of HRV, will be accompanied by the HRV during the techniques and two hours afte
  Interventions: Other: Massage; Other: Exercise

INTERVENTIONS:
Other: Massage — Approximately 12 minutes of massage will be performed in full. The massage will be performed on the lower (anterior) and trunk (posterior)
  Arms: Exercise and Massage after recovery; Exercise and Massage immediately; Only Massage
Other: Exercise — A wingate protocol will be performed followed by 10 sets of 10 squats followed by jumps.
  Arms: Exercise and Massage after recovery; Exercise and Massage immediately; Only Exercise

SUMMARY:
Performing physical exercise alters the body's homeostasis, and recuperative techniques seek to anticipate and potentiate the body's recovery. One of the ways to demonstrate a recovery of the organism is the resumption of autonomic cardiac modulation analyzed through heart rate variability (HRV), a method of global assessment of the behavior of the autonomic nervous system. Among the recovery techniques, massage is the most widely used technique in sports. Therefore, the objective of the study will be to measure the effects of massage as a recuperative technique on autonomic cardiac modulation at different moments of application. It will be a randomized clinical trial where there will be five stages of evaluation. In the first stage, the behavior of the baseline HRV will be evaluated, in the second stage the behavior of the HRV in front of the massage, in the third stage the behavior of the HRV in front of the stress protocol, in the fourth stage the HRV behavior after the stress protocol and immediately after Execution of the massage and finally in the 5th stage where the HRV behavior will be evaluated after the stress protocol and the massage application will be performed at the moment of HRV recovery. The stress protocol will be composed of squats followed by jumps and wingate test, and massage by slides in the anterior thighs and posterior trunk. The HRC indexes in the time domain, frequency domain and Poincaré plot, as well as cardiorespiratory parameters and a questionnaire on individual touch perception will be analyzed. The descriptive statistical method will be used and comparisons of cardiorespiratory parameters and HRV indices will be performed using the analysis of variance technique for repeated measures model in the two factor scheme. The level of significance will be p <0.05 for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Appropriate age limit
* Male

Exclusion Criteria:

* Smokers
* Use of drugs that influence the autonomic modulation of the heart.
* Ethicalists
* Carriers of known metabolic and / or endocrine disorders
* Sedentary individuals, insufficiently active and very active according to IPAQ
* Individuals outside the BMI range

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-09 (Estimated); Primary Completion 2018-05-14 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) - Linear indices - Frequency domain | First 5 minutes of rest; During recovery 5 minutes initial; 10º to 15ºm; 20º to 25ºm; 30º to 35ºm; 40º to 45ºm; 50º to 55ºm; 60º to 65ºm; 70º to 75ºm; 90º to 95ºm; 115º to 120ºm.
  HRV is a noninvasive and selective way of assessing the autonomic function being determined by analyzing the time series of the RR intervals. The HRV analysis will be performed by the Polar Electro Oy - V800 cardiofrequency meter.
  In the analysis of the linear methods, 3 rMSSD, SDNN and pNN50 indices will be used within the time domain. RMSSD corresponds to the square root of the square mean of the differences between the adjacent normal RR intervals in a time interval expressed in milliseconds. The SDNN index represents the standard deviation of all normal RR intervals recorded over a time interval, expressed in milliseconds. And finally, the pNN50 index is the percentage of adjacent RR intervals with a duration difference greater than 50 milliseconds.
Heart Rate Variability (HRV) - Linear indices - Time domain | First 5 minutes of rest; During recovery 5 minutes initial; 10º to 15ºm; 20º to 25ºm; 30º to 35ºm; 40º to 45ºm; 50º to 55ºm; 60º to 65ºm; 70º to 75ºm; 90º to 95ºm; 115º to 120ºm.
  HRV is a noninvasive and selective way of assessing the autonomic function being determined by analyzing the time series of the RR intervals. The HRV analysis will be performed by the Polar Electro Oy - V800 cardiofrequency meter.
  In the analysis of the linear methods, 3 LF, HF and LF / HF indices will be used within the frequency domain. Low frequency corresponds to frequencies between 0.04 and 0.15 Hz (LF - frequency between 0.04 and 0.15 Hz), high frequency (HF - frequency between 0.15 and 0.4 Hz) and the ratio between these components ( LF / HF). These indices shall be expressed in ms² and standard units.
Heart Rate Variability (HRV) - Plot of Poincaré | First 5 minutes of rest; During recovery 5 minutes initial; 10º to 15ºm; 20º to 25ºm; 30º to 35ºm; 40º to 45ºm; 50º to 55ºm; 60º to 65ºm; 70º to 75ºm; 90º to 95ºm; 115º to 120ºm.
  HRV is a noninvasive and selective way of assessing the autonomic function being determined by analyzing the time series of the RR intervals. The HRV analysis will be performed by the Polar Electro Oy - V800 cardiofrequency meter.
  The Poincaré plot is a map of points in Cartesian coordinates constructed from the values of the RR intervals obtained, where each point is represented on the x (horizontal / abscissa) axis by the preceding normal RR interval e, on the y axis (vertical / ordinate) By the following RR interval

SECONDARY OUTCOMES:
Heart rate. | 1, 3, 5, 7, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110 and 120 minutes.
  Heart rate is the number of heartbeats per unit of time. The heart rate will be measured by a heart monitor, and will be displayed in beats per minute (BPM).
Oxygen saturation. | 1, 3, 5, 7, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110 and 120 minutes.
  Oxygen saturation is the percentage of arterial blood hemoglobin that is bound to oxygen. Pulse oximetry will be used to gauge the oxygen saturation, pulse oximetry is the way to measure how much oxygen your blood is carrying. ... The oxygen level measured with a finger oximeter, and the result of this measurement is called the saturation level of oxygen (SatO2)
Respiratory rate. | 1, 3, 5, 7, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110 and 120 minutes.
  Respiratory rate is the designation given to the number of respiratory cycles that is completed in a specific time span, being more commonly expressed in breaths per minute. The respiratory rate will default to 1 minute to express the respiratory cycle number. The respiratory rate will be counted by an evaluator.

CONTACTS AND LOCATIONS:
Locations (1):
- Nilton Mantovani Junior, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mantovani Junior N, Pizzo Junior E, Dos Santos Siqueira M, de Souza Cavina AP, Pastre CM, Marques Vanderlei F. Effects of massage as a recuperative technique on autonomic modulation of heart rate and cardiorespiratory parameters: a study protocol for a randomized clinical trial. Trials. 2018 Aug 25;19(1):459. doi: 10.1186/s13063-018-2830-1. PMID 30144819